CLINICAL TRIAL: NCT00986024
Title: Strength Training Versus Aerobic Interval Training to Modify Risk Factors of the Metabolic Syndrome
Brief Title: Resistance and/or Endurance Training, What is Most Effective in Prevention of Cardiovascular Diseases?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 460150
Record Dates: First submitted 2009-09-28; First posted 2009-09-29 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Metabolic Syndrome
Keywords: Exercise therapy
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- aerobic exercise (Experimental)
  Interventions: Behavioral: aerobic exercise
- strength training (Experimental)
  Interventions: Behavioral: strength training
- control group (No Intervention)

INTERVENTIONS:
Behavioral: aerobic exercise — carried out 3 times per week for 12 weeks
  Arms: aerobic exercise
Behavioral: strength training — carried out 3 times per week for 12 weeks
  Arms: strength training

SUMMARY:
The aim of the present study was to evaluate the effects of aerobic interval training versus strength training or a combination of these regimes on factors comprising the metabolic syndrome in order to find the most effective exercise regime for patients with metabolic syndrome.

DETAILED DESCRIPTION:
In the Western world, approximately 25% of young to middle-aged adults have metabolic syndrome. There seem to be a strong age-dependence in the prevalence of the metabolic syndrome, but the incidence rises rapidly within adolescents and middle-aged groups and follows the development of obesity in the general population. Metabolic syndrome confers an increased risk of coronary heart disease, cardiovascular disease, and premature death; therefore, effective and affordable strategies to combat the syndrome would be of great individual and social importance.

Despite the general agreement that moderate-intensity physical activity for a minimum of 30 min five days per week or vigorous-intensity aerobic physical activity for a minimum of 20 min three days a week promote and maintain health, the optimal training regime to treat metabolic syndrome and its associated cardiovascular abnormalities remains uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Having metabolic syndrome according to international diabetes foundations definition (IDF).

Exclusion Criteria:

* Unstable angina pectoris
* Uncompensated heart failure
* Myocardial infarction during the past 4 weeks
* Complex ventricular arrhythmias
* Kidney failure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
proinflammatory markers | 12 weeks
  circulating interleukin-18 and interleukin-6

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, md prof, Study Director — Norwegian University of Science and Technology

REFERENCES:
- [Result] Stensvold D, Slordahl SA, Wisloff U. Effect of exercise training on inflammation status among people with metabolic syndrome. Metab Syndr Relat Disord. 2012 Aug;10(4):267-72. doi: 10.1089/met.2011.0140. Epub 2012 Mar 28. PMID 22455564